CLINICAL TRIAL: NCT01968174
Title: Astigmatic Corneal Changes Secondary to Eyelid Surgery
Brief Title: Astigmatic Changes Secondary to Eyelid Surgeries
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Meir Medical Center (Other)
Responsible Party: Principal Investigator, shay ofir, SHAY OFIR, Meir Medical Center
Other Study IDs: oculoplasticmeir001
Record Dates: First submitted 2013-10-19; First posted 2013-10-23 (Estimated); Last update posted 2014-08-12 (Estimated); Status verified 2014-08

CONDITIONS: Blepharoptosis
Keywords: astigmatism; lid surgery; older than 40 years; can sign an acceptance form; uper lid surgery
MeSH Terms: conditions — Blepharoptosis; Astigmatism

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 3 Months
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- eyelid displacement: patients suffering from eyelid disposition due to ptosis, blepharochalasis and are registered for eyelid surgeries will be assigned for the study

SUMMARY:
Eyelid surgeries change the lid position over the cornea. Previous surgeries evaluated astigmatic corneal changes in children undergoing ptosis repair. Only several studies evaluated astigmatic changes following eyelid surgeries in elderly patients. The investigators aim is to estimate this change, implications on corneal astigmatism may have great effect to future cataract surgeries for this group of patients.

DETAILED DESCRIPTION:
Patients registered for a lid surgery due to blepharoptosis or ptosis will undergo a topographic examination prior to and 3 months post operative in addition to their regular pre and post operative examination astigmatic shift will be mathematically measured.

ELIGIBILITY:
Inclusion Criteria:

upper lid blepharochalasis

Exclusion Criteria:

prior eyelid trauma mental retardation or other causes preventing from signing an agreement form

Ages: 40 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: patients undergoing eyelid surgery.
Sampling Method: Non-Probability Sample
Enrollment: 30 (Estimated)
Dates: Start 2014-06; Primary Completion 2015-06 (Estimated); Study Completion 2015-06 (Estimated)

PRIMARY OUTCOMES:
astigmatic corneal decrease following eyelid surgery | 3 months
  eyelid change in position will change the effect on corneal astigmatism measured 3 months post surgery

SECONDARY OUTCOMES:
type of astigmatism | 3 months
  a change from against the rule astigmatism to with the rule astigmatism following eyelid surgery will be evaluated

OTHER OUTCOMES:
complications | 3 months
  complications following eyelid surgery and their implications on astigmatism

CONTACTS AND LOCATIONS:
Overall Officials: Arye - Nemet, MD, Principal Investigator — Meir Medical Center
Locations (3):
- Israel (3):
  - Meir Medical center, Kfar Saba, Israel
  - Meir Medical Center, Kfar Saba, Israel
  - Meir Medical Center, Kfar Saba